CLINICAL TRIAL: NCT03911427
Title: Impact of Oat Product on LDL Cholesterol in Healthy Men and Women With Elevated LDL-cholesterol
Brief Title: Oat and Cholesterol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Collaborators: Glycemic Index Laboratories, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PEP-1801
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Elevated LDL Cholesterol
Keywords: Beverage; Beta glucan; Fiber; Oat; Hypercholesterolemia; LDL; Cholesterol
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Gyrate Atrophy; Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Powder Mix 1 (Experimental): Oat powder product, mixed with water
  Interventions: Other: Active oat beverage
- Powder Mix 2 (Placebo Comparator): Brown rice milk powder product, mixed with water
  Interventions: Other: Control rice beverage

INTERVENTIONS:
Other: Active oat beverage — Powder packaged in sachets, mixed with water and consumed 3 times per day for 1 month
  Arms: Powder Mix 1
Other: Control rice beverage — Powder packaged in sachets, mixed with water and consumed 3 times per day for 1 month
  Arms: Powder Mix 2

SUMMARY:
The primary objective is to assess the effect of an oat ingredient provided over 4 weeks on serum LDL cholesterol in men and women with elevated LDL-cholesterol compared to a placebo.

Secondary endpoints are fasting serum total- and HDL-cholesterol, non-HDL-cholesterol, triglycerides, glucose, insulin, glycated albumin, HOMA-IR and Framingham risk score

ELIGIBILITY:
Inclusion Criteria:

1. Fasting LDL cholesterol 116-193 mg/dl (3-5 mmol/L)
2. Males and non-pregnant, non-lactating females 18-65 years
3. Agree to consume the investigational product three times daily for the duration of the study
4. BMI 18.5 to 39.9 kg/m2
5. Blood pressure <160/100 mmHg
6. Fasting triglycerides <4.0 mmol/L
7. Fasting serum glucose <126mg/dL (<7 mmol/L)
8. Serum urea and creatinine < 1.8 times upper limit of normal (ULN)
9. Serum aspartate aminotransaminase (AST), alanine aminotransferase (ALT) and gamma-glutamyl transferase (GGT) < 2 times ULN
10. Hemoglobin > 0.9 times lower limit of normal and < 1.1 times ULN
11. Have a stable body weight (<7 kg change) over the past 3-months
12. Absence of health conditions that would prevent fulfillment of study requirements

Exclusion Criteria:

1. Pregnancy, breastfeeding or planning to be pregnant
2. Allergy or sensitivity to study product ingredients
3. Dislike description of study product
4. Diet containing ≥15% of energy from saturated fat
5. Consuming >20g fiber/per 1000 Kcal or >40g fiber/day (including soluble fiber supplements)
6. Consumption of more than 2 drinks of alcohol per day, or more than 14 drinks per week
7. Extreme dietary habits
8. Smoking >5 cigarettes or equivalent per day
9. Use of cholesterol lowering medication or prescription drug or for treating diabetes mellitus within 4 weeks of randomization
10. Active major gastrointestinal disorder
11. Major trauma or hospitalization for a medical condition or major surgical event within 6 months of randomization
12. History of cancer within two years or randomization, except for non-melanoma skin cancer
13. Any condition or substance use which might, in the opinion of the PI, make participation dangerous for the participant, lead to poor attendance or compliance or affect the results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Change in fasting serum LDL-cholesterol | Baseline vs. Week 4
  Reduction in mmol/L is a better outcome and >=5% reduction would be significant

SECONDARY OUTCOMES:
Change in fasting serum total cholesterol | Baseline vs. Week 4
  Reduction in mmol/L is a better outcome
Change in fasting serum HDL cholesterol | Baseline vs. Week 4
  Increase in mmol/L is a better outcome
Change in fasting non-HDL-cholesterol | Baseline vs. Week 4
  Reduction in mmol/L is a better outcome
Change in fasting triglycerides | Baseline vs. Week 4
  Reduction in mmol/L is a better outcome
Change in fasting glucose | Baseline vs. Week 4
  Reduction in mmol/L is a better outcome
Change in fasting insulin | Baseline vs. Week 4
  Reduction in mmol/L is a better outcome
Change in fasting glycated albumin | Baseline vs. Week 4
  % reduction is a better outcome. Normal range is 11-17% of total albumin.
Change in fasting HOMA-IR | Baseline vs. Week 4
  Reduction is a better outcome. Calculated from serum glucose mmol/L and insulin uU/ml. G×I/22.5, where G is fasting serum glucose in mmol/L and I is fasting serum insulin in uU/mL. Less than 1.0 means insulin-sensitive, which is optimal. Above 1.9 indicates early insulin resistance. Above 2.9 indicates significant insulin resistance.
Change in Framingham risk score | Baseline vs. Week 4
  Reduction is a better outcome. 10 year risk for cardiovascular disease = total points expressed as % for men and women. Calculated from sex, age, total and HDL cholesterol (mg/dL), systolic blood pressure (mmHg), smoking (yes/no) and diabetes (yes/no) using the equations given on the Framingham Heart Study website.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas MS Wolever, MD, PhD, Principal Investigator — Glycemic Index Laboratories, Inc
Locations (1):
- Glycemic Index Laboratories, Inc. 20 Victoria Street, 3rd Floor, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ms Wolever T, Rahn M, Dioum E, Spruill SE, Ezatagha A, Campbell JE, Jenkins AL, Chu Y. An Oat beta-Glucan Beverage Reduces LDL Cholesterol and Cardiovascular Disease Risk in Men and Women with Borderline High Cholesterol: A Double-Blind, Randomized, Controlled Clinical Trial. J Nutr. 2021 Sep 4;151(9):2655-2666. doi: 10.1093/jn/nxab154. PMID 34236436